CLINICAL TRIAL: NCT03839862
Title: Faecal Analyses in Spondyloarthritis Therapy: A Prospective Observational Study of the Intestinal Microbiome in Patients With Spondyloarthropathy Receiving TNF-inhibition.
Brief Title: Faecal Analyses in Spondyloarthritis Therapy
Acronym: FAST
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: FAST1
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Spondyloarthropathies; Ankylosing Spondylitis
MeSH Terms: conditions — Spondylarthropathies; Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and faecal sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Responder: Patient responding to TNF-inhibition
  Interventions: Drug: TNF-inhibition
- non-Responder: Patient not responding to TNF-inhibition
  Interventions: Drug: TNF-inhibition

INTERVENTIONS:
Drug: TNF-inhibition — Initiation of immunosuppression with any TNF-inhibitor, e.g. infliximab, etanercept or adalimumab

SUMMARY:
This study evaluates the intestinal microbiome and disease activity in patients with spondyloarthropathies receiving immunosuppressive therapy.

Patients will be analysed at two time points in reference to two predefined primary endpoints:

* Changes in intestinal microbiome
* Response to therapy

The investigators want to evaluate if successful treatment of spondylarthropathy coincide with specific changes in the gut flora.

DETAILED DESCRIPTION:
Tumor necrosis factor (TNF)-inhibition is an efficient medication for the treatment of spondyloarthropathy. In a substantial number of cases however, these medications remain ineffective. At present, the scientific community has limited understanding of why some patients are resistant to this medication. The purpose of this study is to understand if the gut flora may associate with treatment response.

Spondyloarthropathies are associated with inflammatory bowel diseases in terms of epidemiology and molecular pathogenesis. Recent studies have also associated spondyloarthropathies with intestinal dysbiosis.

This study is of observational character and integrated in the routine clinical care of patients with spondyloarthropathies at the Rheumatology Clinic, Skane University Hospital, Lund, Sweden. Study participants are asked to deliver blood and fecal sampling at two time-points together with clinical evaluation of disease activity. With an estimated inclusion of 50 patients, at least 20 responders and 20 non-responders are expected to be included and to be compared to each other.

Our primary goal is to investigate the association between change in intestinal microbiome and clinical response to therapy.

In our secondary analyses we will investigate if intestinal microbiome and intestinal inflammation at baseline may predict response to, and adherence to, therapy in these patients.

If successful treatment response of spondyloarthropathy is associated with specific alterations of the gut flora, these results may guide future studies on the impact of dysbiosis and probiotics on this disease.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling the Assessment of SpondyloArthritis International Society classification criteria for spondyloarthropathy.
* About to commence treatment with TNF-inhibition

Exclusion Criteria:

* Failure to understand protocol
* A history of alcohol abuse
* Any history of diverticulitis
* A history of failure to comply with prescribed medication
* Ongoing biological therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study encompasses consecutive patients with spondyloarthropathy who by their physician at the Rheumatology Clinic, Skåne University Hospital, have been prescribed a TNF-inhibitor.
  Patients who are willing to comply with the study protocoll are included. The study population is consequently not a sample, but encompasses a majority of spondyloarthropathy patients being prescribed this medication at our University clinic.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in gut flora | Change from baseline Dysbiosis Index Score at 6 months
  Change in Dysbiosis Index Score att follow up compared to baseline. The Dysbiosis Index Score measures degree of intestinal dysbiosis on a scale from 1 to 5, where 5 indicates dysbiosis.
Change in disease activity/treatment response at follow up | Change from baseline BASDAI at 6 months
  Change in Bath Ankylosing Spondylitis Disease Activity Score (BASDAI), an established index of disease activity in spondylarthropathies between 0-10, where 10 equals maximum activity

SECONDARY OUTCOMES:
Intestinal gut flora in spondyloarthropathies | Analysis made at study start /baseline
  Intestinal gut flora based on DNA-based microbial analysis of fecal samples (Dysbiosis Index Score). The Dysbiosis Index Score measures degree of intestinal dysbiosis on a scale from 1 to 5, where 5 indicates dysbiosis.
Intestinal gut inflammation | Analysis made at study start /baseline
  Assessment of intestinal inflammation by measurement of faecal calprotectin, an established biomarker of intestinal inflammation
Adherence to immunosuppressive therapy | Analysis made at 6 months follow up
  Is the patient still prescribed the same immunosuppressant compared to baseline?

CONTACTS AND LOCATIONS:
Overall Officials: Kristofer Andréasson, MD PhD, Principal Investigator — Lund University Hospital
Locations (1):
- Reumatologi SUS Lund, Region Skåne, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No